CLINICAL TRIAL: NCT06075056
Title: Neuro-navigated TMS for Chronic SCI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: King's College Hospital
Record Dates: First submitted 2023-01-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic spinal cord injuries: Defined as spinal cord injuries secondary to a single traumatic event to the Cervical or thoracic spine, more than 6 months ago.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention is planned as part of this study, this is a feasibility/pilot study

SUMMARY:
Can neuro-navigated Transcranial Magnetic Stimulation be used as an additional outcome measure to EM-SCI assessments in a Spinal cord injury trial?

* Compare EM-SCI assessment with nTMS in ten chronic thoracic SCI patients
* Compare EM-SCI assessment with nTMS in ten chronic cervical SCI patients

DETAILED DESCRIPTION:
This is an exciting time for translating experimental Advanced Therapies into treatments for spinal cord injury (SCI). There are currently no regenerative therapies available that target the underlying biology. Over the last 5 years the investigating team have developed a viable gene therapy approach for treating SCI in pre-clinical models. The investigators are on the cusp of translating this therapy to first-in-human studies and are leading a programme to establish a world-first regenerative gene therapy for traumatic SCI affecting upper limb mobility (since recovery of arm/hand function is one of the highest patient priorities). The team will develop an innovative trial design involving neurosurgical delivery of the gene therapy into the spinal cord, followed by specialist neurorehabilitation.

For a clinical trial to have the best chance of success, one of the key steps needed to be addressed include validation of new assessment methods for the clinical trial. Our aim is to determine whether neuro-navigated Transcranial Magnetic Stimulation (nTMS) can be used as an adjunct to standard assessments of function in SCI patients. Following two patient and public involvement events (patient focus group and feedback for project design with our rehabilitation partners), the investigating team will recruit chronic SCI subjects to carry out European Multicenter Study about SCI (EM-SCI) assessments. EM-SCI assessments are well established assessment tools for SCI patients and include the EM-SCI 'core' assessments (ISNCSCI, WISCI-III, Walk Test, SCIM 3) and EM-SCI 'additional' assessments (GRASSP, Pain score, neurophysiology). Following this investigators will compare and validate nTMS with EM-SCI assessments in stable chronic SCI patients with both cervical and thoracic injuries. nTMS with combined Tractography MRI of the cortico-spinal tract (the main motor pathway of the spinal cord) will allow functional characterisation and density measurements of this tract in SCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Single traumatic event at least 6 months prior to recruitment
* ISNCSCI grade A, B, C or D
* Able to participate in EM-SCI and nTMS assessments and capable of informed consent

Exclusion Criteria:

* History of Malignancy
* History of other Neurological disease
* Pregnancy
* Other cord lesions or tethering
* Cord transaction or penetrating injury

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 20 patients, 10 Cervical SCI and 10 Thoracic SCI who meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Resting Motor Threshold (rMT) | 1 year
  Resting motor threshold (rMT) is the amount of machine output responsible for a positive motor evoked potential in at least % of the trials. This outcome is expressed in % and it is directly obtained from the TMS software.
Motor Evoked Potential (MEP) Latency | 1 year
  MEP latency is a TMS measure of time taken for intracortical processing, spinal processing and neurmuscular transmission. It is measure in miliseconds (mS). Linear regression analysis will be used to compare TMS measurements against EM-SCI measurements to validate TMS as an assessment tool for chronic SCI.
Motor Evoked Potential (MEP) amplitude | 1 year
  Motor evoked potential (MEP) Amplitude is a TMS measurement of the number of motoneurons recruited during TMS stimulation. It is expressed in milivolt (mV). Linear regression analysis will be used to compare TMS measurements against EM-SCI measurements to validate TMS as an assessment tool for chronic SCI.
Spinal cord independence measure III (SCIM III) | 1 year
  SCIM is a validated reproducible measure used in EM-SCI, as a measure of spinal cord injury functionality. This is a questionnaire with a score from 0-100.
Graded redefined assessment of strength, sensation and prehension (GRASSP) | 1 year
  GRASSP is a validated clinical impairment score to measure impairment in the upper limbs. This is a tool currently used within the EM-SCI protocol.
Diffusion Tension Imaging Metrics of Corticospinal Tract Tractography | 1 year
  We will calculate the fractional anisotropy, radial diffusivity, axial diffusivity and mean diffusivity for bilateral cortical spinal tract. These metrics range from 0 to 1. We will use DSI Studio Software to proceed with these calculations.
Cortical Motor Area and Volume | 1 year
  We will calculate the area and volume of cortical activation of both upper and lower limbs.The area is calculated in cm2 and the volume in microvolt per cm2. We will use TMSMap Software to produce these metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Aminul Ahmed, Principal Investigator — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT06075056/Prot_000.pdf
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT06075056/ICF_001.pdf